CLINICAL TRIAL: NCT05809466
Title: The Effect of a 12-week Self-composed Vegan Diet With or Without Concurrent Resistance Exercise on Thigh Muscle Volume in Older Adults
Acronym: Vold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Lisette de Groot, Prof. Dr. Ir. L.C.P.G.M. (Lisette) de Groot, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL82788.091.22
Record Dates: First submitted 2023-03-14; First posted 2023-04-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-11

CONDITIONS: Vegan Diet; Sarcopenia; Cardiovascular Health; Osteoporosis; Gut Health
MeSH Terms: conditions — Sarcopenia; Osteoporosis | interventions — Diet, Vegan; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vegan group (Experimental)
  Interventions: Other: Vegan diet
- Vegan group with resistance exercise (Experimental)
  Interventions: Other: Vegan diet; Other: Resistance exercise
- Omnivorous group (Active Comparator)
  Interventions: Other: Omnivorous diet

INTERVENTIONS:
Other: Vegan diet — A self-composed 12 week fully plant-based diet
  Arms: Vegan group; Vegan group with resistance exercise
Other: Resistance exercise — Biweekly resistance exercise for 12 weeks
  Arms: Vegan group with resistance exercise
Other: Omnivorous diet — Habitual diet containing both animal- and plant-based food products
  Arms: Omnivorous group

SUMMARY:
Consumers are increasingly encouraged to consume more plant-based foods and lower their consumption of foods from animal origin. This shift is driven by environmental and health factors. However, the consequences of such a transition on muscle mass still remains to be explored. This is of particular importance in the older population, where the age-related reduction in muscle mass and strength is highly prevalent. Adequate dietary intake, specifically protein intake, is a well-known strategy in promoting muscle mass in older adults. Plant-based foods are currently considered to be inferior to animal-based foods in their protein quality, and are therefore considered to be suboptimal for the maintenance of muscle mass at an older age. On the other hand, combining plant-based foods may improve the protein quality and thereby the anabolic properties of a vegan meal. Evidence regarding the anabolic properties of vegan diets in older adults is scarce. As such, the current study aims to assess 1) the effects of a 12-week self-composed vegan diet in comparison to an omnivorous diet on thigh muscle volume (TMV) in community-dwelling older adults and 2) the effect of a 12-week self-composed vegan diet combined with twice-weekly resistance exercise (RE) on TMV in comparison to a self-composed vegan diet without resistance exercise in community-dwelling older adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥65 years old;
* Community-dwelling;
* BMI 23-32 kg/m2;
* Habitual diet contains animal-based food products (i.e. dairy, meat and/or fish) at least 5 days per week;

Exclusion Criteria:

* Following a self-reported entirely vegetarian or vegan diet during the six months prior to the study;
* Following a prescribed high (≥1.2 g/kg/d) or low protein diet (<0.8 g/kg/d), and/or or taking protein supplements on medical advice, during the month prior to the study;
* Participating in a structured progressive resistance exercise training program the during three months prior to the study;
* ≥4 kg of body weight loss during three months before the start of the study;
* Being diagnosed with one of the following: diabetes mellitus; renal disease; neurological or neuromuscular disorders; serious cardiovascular diseases; cancer (with the exception of the following types of skin cancer: basal cell carcinoma, squamous cell carcinoma); (very) severe chronic obstructive lung disease (COPD; GOLD stage III or IV); bowel disease.
* Chronic use of medication that affects muscle function as assessed by the research physician;
* The use of anticoagulants incompatible for muscle biopsies as assessed by the research physician: acenocoumarol (sintrom); phenprocoumon (marcoumar); dabigatran (pradaxa); apixaban (eliquis); rivaroxaban (xarelto); clopidogrel (plavix); edoxaban (lixiana); combination of acetylsalicylic acid or carbasalate calcium (ascal) with dipyridamole;
* Having a contra-indication to MRI scanning (including, but not limited to):

  * Pacemakers and defibrillators
  * Infraorbital or intraocular metallic fragments
  * Ferromagnetic implants
  * Claustrophobia
* Having a hip prosthesis
* Not willing to stop nutritional supplements, with the exception of supplements on medical advice, and vitamin D;
* Not willing or afraid to give blood, undergo a muscle biopsy or have an MRI scan during the study;
* Unwilling to eat a self-composed vegan diet or an omnivorous diet with daily consumption of animal-based food sources for 3 months;
* Unwilling to participate in RE twice a week for 3 months;
* Currently a research participant in another trial or participated in a clinical trial during one month before the start of the measurement period;
* Not being able to understand Dutch;
* Not having a general physician;
* Working, or having a direct family member that work at the Division of Human Nutrition at Wageningen University during the study.
* Unwilling to be informed about incidental findings of pathology and approving of reporting this to their general physician.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Change in thigh muscle volume | 12 weeks
  Thigh muscle volume of both legs will be assessed using magnetic resonance imaging before and after the 3-month intervention

SECONDARY OUTCOMES:
Body composition | Change after 12 weeks
  Other body composition indices will also be measured using magnetic resonance imaging before and after the intervention. These indices include: liver fat fraction, thigh muscle fat infiltration, abdominal subcutaneous adipose tissue, visceral fat tissue.
Change in muscle strength | Change after 12 weeks
  Maximal isometric knee extension and flexion strength of both legs will be measured using Biodex.
Muscle fractional synthesis rates | 10 days
  Muscle fractional synthesis rates, expressed as daily fractional synthesis rates (FSR, %/day), will be assessed using a deuterium oxide protocol. Daily FSR will be calculated using the 2^H-alanine enrichment in plasma and the mixed muscle-bound 2^H-alanine enrichment.
Change in bone mineral density | Change after 12 weeks
  Measured using a Dual X-Ray Absorptiometry dual femur scan
Change in fasting bone turnover markers | Change after 6 and 12 weeks
  Serum procollagen type I N-terminal propeptide (P1NP) will be measured for bone formation and C-terminal telopeptide of type I collagen (CTX) for bone resorption.
Change in plasma insulin growth factor 1 levels | Change after 6 and 12 weeks
  Fasting serum insulin-like growth factor 1 (IGF-1)
Change in plasma parathyroid hormone (PTH) levels | Change after 6 and 12 weeks
  Fasting plasma PTH
Change in fasting plasma insulin levels | Change after 6 and 12 weeks
  Fasting plasma insulin
Change in metabolic profile | Change after 6 and 12 weeks
  Fasting plasma levels of multiple metabolites
Change in fasting blood pressure | Change after 6 and 12 weeks
  Fasting systolic and diastolic blood pressure
Change in haemoglobin levels | Change after 12 weeks
  Fasting plasma haemoglobin levels
Change in vitamin B12 status | Change after 12 weeks
  Fasting plasma methylmalonic acid levels
Change in vitamin D status | Change after 12 weeks
  Fasting serum vitamin D levels
Change in gastro-intestinal symptoms | Change after 12 weeks
  Self-reported gastro-intestinal symptoms using the gastro-intestinal symptom rating scale. The questionnaire includes 15 questions covering 5 common symptom clusters on a 7-point likert scale ranging from no symptoms (minimum) to severe symptoms (maximum). A higher score indicates worse symptoms.
Untargeted gut metabolomics | Change after 12 weeks
  Untargeted gut metabolomics will be performed on fasting plasma samples
Change in fasting plasma high-sensitive C-reactive protein (hs-CRP) | Change after 6 and 12 weeks
  Fasting plasma hs-CRP
Change in ferritin levels | Change after 12 weeks
  Fasting plasma ferritin levels
Tryptophan | Change after 12 weeks
  Tryptophan will be assessed using targeted metabolomics on plasma samples
Tyrosine | Change after 12 weeks
  Tyrosine will be assessed using targeted metabolomics on plasma samples
Branch-chained amino acids | Change after 12 weeks
  Branch-chained amino acids will be assessed using targeted metabolomics on plasma samples
Oxidized amino acids | Change after 12 weeks
  Oxidized amino acids will be assessed using targeted metabolomics on plasma samples
Gut metagenomics | Change after 12 weeks
  Microbial DNA will be isolated from the feces samples. The taxonomy and function of specific genes will be assessed via metagenomic sequencing on the microbial DNA.

OTHER OUTCOMES:
Change in body weight | Change after 10 days and after 12 weeks
  Body weight (kg) will be measured in a fasted state using a calibrated digital scale

CONTACTS AND LOCATIONS:
Overall Officials: Lisette de Groot, PhD, Principal Investigator — Wageningen University and Research
Locations (1):
- Wageningen University and Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Domic J, Grootswagers P, Pinckaers PJ, Groenendijk I, Rubert J, van Loon LJ, de Groot LC. The effect of a vegan diet with or without resistance exercise on thigh muscle volume in older adults. Research protocol of the Vold-study: a 12-week randomized controlled trial. BMC Geriatr. 2025 Dec 26;26(1):120. doi: 10.1186/s12877-025-06708-9. PMID 41454225